CLINICAL TRIAL: NCT06975501
Title: A Community-Based 2×2 Factorial Randomized Controlled Trial Evaluating a Multicomponent Physical and Cognitive Intervention for Older Adults With Stroke and Comorbid Chronic Conditions in Urban China
Brief Title: Community-Empowerment and Environmental Enrichment-based Co-management (CEEEC) Model and Mechanisms for Improving Health of Older Stroke Patients With Multimorbidity
Acronym: CEEEC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke Kunshan University (Other)
Collaborators: Wuhan University (Other); Harbin Medical University (Other); Shanghai Jiao Tong University School of Medicine (Other); Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Lijing Yan, Professor, Duke Kunshan University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025DKU
Record Dates: First submitted 2025-04-30; First posted 2025-05-16 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-05

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus (T2DM); Multimorbidity; Stroke
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Control (No Intervention): Participants in this arm will receive medication compliance education from the family doctor.
- Physical Activity Only (Experimental): Participants will receive twice-weekly aerobic and balance training sessions, with medication compliance education.
  Interventions: Behavioral: Exercise Intervention
- Cognitive Training Only (Experimental): Participants in this arm will participate in twice-weekly structured cognitive training sessions, with medication compliance education.
  Interventions: Behavioral: Cognitive Intervention
- Combined Physical + Cognitive (Experimental): Participants in this arm will receive both twice-weekly aerobic and balance training sessions and twice-weekly structured cognitive training sessions, with medication compliance education.
  Interventions: Behavioral: Exercise Intervention; Behavioral: Cognitive Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention — Participants will receive twice-weekly aerobic and balance training sessions, with medication compliance education.
  Arms: Combined Physical + Cognitive; Physical Activity Only
Behavioral: Cognitive Intervention — Participants will participate in twice-weekly structured cognitive training sessions, with medication compliance education.
  Arms: Cognitive Training Only; Combined Physical + Cognitive

SUMMARY:
This study is a cluster randomized controlled trial with a 2×2 factorial design conducted in community health centers in Kunshan, Harbin, Wuhan, Beijing and Shanghai. It aims to evaluate the independent and combined effects of exercise and cognitive interventions on intrinsic capacity and related health outcomes among stroke survivors aged 60 years and older with hypertension or type 2 diabetes mellitus. Participants will receive either exercise training, cognitive training, combined training, or usual care over 12 months, followed by a 12-month follow-up. Findings will inform integrated health management strategies for older adults with multimorbidity.

DETAILED DESCRIPTION:
This study is a community-based cluster randomized controlled trial with a 2×2 factorial design, conducted in community health centers in Kunshan (Jiangsu), Wuhan (Hubei), Harbin (Heilongjiang), Beijing and Shanghai, China. A total of 480 stroke survivors aged 60 years and above with comorbid hypertension or type 2 diabetes mellitus will be recruited. Participants will be randomly assigned to one of four groups: exercise intervention only, cognitive intervention only, combined intervention, or control (usual care). The interventions, including aerobic-balance physical training and structured cognitive training, will be delivered twice weekly for 12 months, followed by a 12-month observational follow-up.

The primary outcome is intrinsic capacity (IC), assessed using the World Health Organization Integrated Care for Older People (WHO ICOPE) framework. Secondary outcomes include systolic blood pressure, quality of life (EuroQol 5-Dimension 5-Level, EQ-5D-5L), medication adherence, physical activity (Metabolic Equivalent of Task minutes per week, MET-min/week), and healthcare utilization. Data will be collected at baseline, 6, 12, and 24 months.

Intervention effects and trajectories over time will be analyzed using two-way analysis of variance (ANOVA), repeated measures ANOVA, and mixed-effects models. Implementation outcomes will be evaluated following the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework. The study aims to generate evidence for integrated health management strategies for older adults with stroke and multimorbidity in urban China.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥60 years
* The doctor diagnosed it as a stroke and it is in a stable stage (the diagnosis time is not limited)
* Patients with concurrent hypertension and/or diabetes may also have other diseases at the same time
* Be able to participate in a community intervention lasting for six months
* Be informed and agree to participate in the research

Exclusion Criteria:

* With the aid of a walking aid (not a wheelchair), it is also impossible to walk independently to the community service center.
* Lack basic communication skills and do not recognize Arabic numerals
* Suffering from life-threatening diseases, with a survival expectation of less than 6 months, etc.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Intrinsic Capacity (World Health Organization Integrated Care for Older People) | 24 months
  Assessment of intrinsic capacity using the World Health Organization Integrated Care for Older People (WHO ICOPE) framework.

SECONDARY OUTCOMES:
Locomotion: SPPB (Short Physical Performance Battery) | 24 months
  The Short Physical Performance Battery (SPPB) is a validated, performance-based tool designed to assess lower extremity function in older adults. It consists of three components: a balance test, a gait speed test, and a chair stand test. Each component is scored on a scale from 0 to 4, with a total score ranging from 0 (worst performance) to 12 (best performance).
Cognition | 24 months
  Cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a widely validated screening tool for mild cognitive impairment. The MoCA evaluates multiple cognitive domains, including attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
  The MoCA score ranges from 0 to 30, with higher scores indicating better cognitive function. A score of 26 or above is generally considered within the normal range.
  Assessments will be conducted at baseline and at regular intervals across the 24-month study period to track changes over time.
Psychological well-being | 24 months
  Psychological well-being will be assessed using the Cornell Scale for Depression in Dementia (CSDD), a clinician-administered instrument specifically designed to assess signs of depression in individuals with cognitive impairment, including those with dementia. The CSDD incorporates information from both patient interviews and caregiver reports to increase the reliability of the assessment.
  The scale includes 19 items, each scored from 0 (absent) to 2 (severe), resulting in a total score ranging from 0 to 38. Higher scores indicate more severe depressive symptoms, reflecting poorer psychological well-being. A score of ≥12 suggests probable major depression, while scores between 8-11 indicate possible depression.
  CSDD assessments will be performed at baseline and repeated at regular intervals throughout the 24-month study period.
Vitality | 24 months
  Vitality will be assessed using the Mini Nutritional Assessment (MNA), a validated screening and assessment tool designed to identify older adults at risk of malnutrition or undernutrition, which are closely associated with reduced physical vitality and frailty.
  The full MNA consists of 18 items, producing a total score ranging from 0 to 30. Higher scores indicate better nutritional status, reflecting greater vitality and overall health.
  A score of 24-30 indicates normal nutritional status. Scores 17-23.5 suggest risk of malnutrition. Scores <17 indicate malnutrition. The MNA will be administered at baseline and at regular follow-ups over the 24-month study period to monitor changes in patients' nutritional status and associated vitality.
Medication Adherence | 24 months
  measured using the 4-item Morisky Green Levine Scale-4 (MMAS-4). The 4-item Morisky Green Levine Medication Adherence Scale (MMAS-4), is a validated self-reported questionnaire that evaluates patients' behaviors related to medication-taking. The scale consists of 4 yes/no questions, with each "yes" answer scored as 1 and each "no" as 0. The total score ranges from 0 to 4, with higher scores indicating lower adherence.
  A score of 0 indicates high adherence. 1-2 indicates medium adherence. 3-4 indicates low adherence.
Physical Activity (MET-min/week) | 24 months
  Measurement of physical activity levels in metabolic equivalent of task (MET) minutes per week.
Systolic Blood Pressure (SBP) | 24 months
  Change in the systolic blood pressure.
Weight | 24 months
  change in weight
Height | 24 months
  change in height
Neck circumference | 24 months
  participants' neck circumference
Waist circumference | 24 months
  Participants' waist circumference
Mobility | 24 months
  measured by timed-up-and-go test, a simple and quick functional mobility test that requires the participants to stand up, walk 3 meters, turn, walk back, and sit down
Mental Health | 24 months
  The Geriatric Depression Scale - 15 item version (GDS-15) is a self-report questionnaire designed to screen for depression in older adults. It contains 15 yes/no questions that assess mood, motivation, energy levels, and outlook on life over the past week. Scores range from 0 to 15, with higher scores indicating more severe depressive symptoms, thus reflecting a worse outcome. Each depressive answer is scored as 1 point, and the total score is the sum of these points. Commonly used cut-off points are: 0-4 (no depression), 5-8 (mild depression), 9-11 (moderate depression), and 12-15 (severe depression).
Health related quality of life | 24 months
  measured using EuroQol-5 Dimensions-5L (EQ5D-5L). EQ-5D-5L descriptive system comprises the following five dimensions, each describing a different aspect of health: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. For each domain, the total scores range from 0 (indicating no problem) to 5 (indicating unable to/extreme problems). In addition, the participants were required to assess how their health is today by write a number from 0 to 100 on the numbered scale. 100 means the best health the participant can image, 0 means the worst health the participant can image.
Lifestyle risk factors | 24 months
  The factors include lack of exercise, alcohol, diet, obesity, and smoking, and will be collected through questionnaire.
Basic activities of daily living | 24 months
  measured by the basic activities of daily living (ADL). The basic ADL include the following categories: Ambulating, Feeding, Dressing, Personal hygiene, Continence, and Toileting. The ADL score ranges from 0 to 12. Limitation in ADL was defined as being scored greater than 0 on ADL scales, i.e., having some or severe limitation in at least one ADL item. Higher scores mean a worse functional independence.
Instrumental activities of daily living | 24 months
  measured by the Lawton Instrumental Activities of Daily Living (IADL) Scale to evaluate independent living skills. The scale measures eight domains of function, including food preparation, housekeeping, laundering. The IADL score ranges from 0 to 14. Limitation in IADL was defined as being scored greater than 0 on IADL scales, i.e., having some or severe limitation in at least one IADL item. Higher scores mean a worse functional independence.
Disability | 24 months
  measured using modified Rankin Scale (ranged 0 (no symptom) to 5 severe disability)
Multimorbidity | 24 months
  Assessed by determining whether participants had additional diseases diagnosed in the hospital, excluding stroke
Locomotion: Grip strength | 24 months
  Grip strength (kilogram) will be estimated through the dynamometer (YuejianTM WL-1000, Nantong, China). Trained examiners will instruct people to hold the dynamometer and squeeze the handle for a few seconds. This study both measures right and left-hand grip strength twice in each hand. The grip strength will be recorded separately. If the average grip strength of both right and left hand of is all less than the criteria (man < 30 kg, woman < 20 kg), it is defined as weak grip strength.
Continuation of medication taking | 24 months
  Measured by the total number of months during the 24-month follow-up period that the patient continuously takes the prescribed medication.
Healthcare Utilization: Hospital Visits | 24 months
  The number of hospital visits (both inpatient and outpatient) will be measured during the 24-month follow-up period. This will include the total number of hospital admissions, along with any follow-up outpatient visits associated with hospital care. Unit of Measure: Number of hospital visits
Healthcare Utilization: Emergency Room Visits | 24 months
  The number of emergency room visits will be assessed over the 24-month period. This includes any visits to the emergency room for acute health concerns or urgent care needs.
  Unit of Measure: Number of emergency room visits
Healthcare Utilization: Outpatient Visits | 24 months
  The number of outpatient visits (excluding emergency room and inpatient visits) will be measured throughout the 24-month study period. This includes visits to primary care providers, specialists, and other outpatient services.
  Unit of Measure: Number of outpatient visits
Self-reported disease history (via questionnaire) | 24 months
  Presence of chronic diseases reported by participants through a structured questionnaire. Unit of Measure: Count of documented diseases
Disease history based on medical insurance records | 24 months
  Number and type of diagnosed chronic diseases retrieved from participants' medical insurance claims data. Unit of Measure: Count of documented diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Kunshan University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The investigators will not share the individual participant data. But de-identified data is available upon request.

REFERENCES:
- [Result] Ni Z, Atluri N, Shaw RJ, Tan J, Khan K, Merk H, Ge Y, Shrestha S, Shrestha A, Vasudevan L, Karmacharya B, Yan LL. Correction: Evaluating the Feasibility and Acceptability of a Mobile Health-Based Female Community Health Volunteer Program for Hypertension Control in Rural Nepal: Cross-Sectional Study. JMIR Mhealth Uhealth. 2020 Jun 11;8(6):e19048. doi: 10.2196/19048. PMID 32525811
- [Result] Gong E, Lu H, Shao S, Tao X, Peoples N, Kohrt BA, Xiong S, Kyobutungi C, Haregu TN, Khayeka-Wandabwa C, Van Minh H, Hanh TTD, Koirala S, Gautam K, Yan LL. Feasibility assessment of invigorating grassrooTs primary healthcare for prevention and management of cardiometabolic diseases in resource-limited settings in China, Kenya, Nepal, Vietnam (the FAITH study): rationale and design. Glob Health Res Policy. 2019 Nov 12;4:33. doi: 10.1186/s41256-019-0124-0. eCollection 2019. PMID 31742234
- [Result] Yan LL, Gong E, Gu W, Turner EL, Gallis JA, Zhou Y, Li Z, McCormack KE, Xu LQ, Bettger JP, Tang S, Wang Y, Oldenburg B. Effectiveness of a primary care-based integrated mobile health intervention for stroke management in rural China (SINEMA): A cluster-randomized controlled trial. PLoS Med. 2021 Apr 28;18(4):e1003582. doi: 10.1371/journal.pmed.1003582. eCollection 2021 Apr. PMID 33909607
- [Result] Tian M, Ajay VS, Dunzhu D, Hameed SS, Li X, Liu Z, Li C, Chen H, Cho K, Li R, Zhao X, Jindal D, Rawal I, Ali MK, Peterson ED, Ji J, Amarchand R, Krishnan A, Tandon N, Xu LQ, Wu Y, Prabhakaran D, Yan LL. A Cluster-Randomized, Controlled Trial of a Simplified Multifaceted Management Program for Individuals at High Cardiovascular Risk (SimCard Trial) in Rural Tibet, China, and Haryana, India. Circulation. 2015 Sep 1;132(9):815-24. doi: 10.1161/CIRCULATIONAHA.115.015373. Epub 2015 Jul 17. PMID 26187183
- [Result] Yan LL, Fang W, Delong E, Neal B, Peterson ED, Huang Y, Sun N, Yao C, Li X, MacMahon S, Wu Y. Population impact of a high cardiovascular risk management program delivered by village doctors in rural China: design and rationale of a large, cluster-randomized controlled trial. BMC Public Health. 2014 Apr 11;14:345. doi: 10.1186/1471-2458-14-345. PMID 24721435
- [Result] Zhu G, Malhotra R, Xiong S, Chen X, Zhang M, Wu Y, Gong E, Wang Z, Tian X, Peng W, Ostbye T, Yan LL. Community Efficacy for Non-Communicable Disease Management and Medication Adherence: The Sequential Mediating Role of Self-Efficacy and Depressive Symptoms. Patient Prefer Adherence. 2023 Dec 14;17:3421-3433. doi: 10.2147/PPA.S436419. eCollection 2023. PMID 38111691
- [Result] Xiong S, Zhu G, Malhotra R, Chen X, Gong E, Wang Z, Zhang J, Peng W, Wang S, Jin X, Peoples N, Ostbye T, Tian M, Yan LL. Community efficacy for non-communicable disease management (COEN): Conceptualization and measurement. PLOS Glob Public Health. 2024 Aug 14;4(8):e0003549. doi: 10.1371/journal.pgph.0003549. eCollection 2024. PMID 39141640